CLINICAL TRIAL: NCT03631459
Title: Safety and Effectiveness of Kanglaite Injection/Capsules for Treatment of Cancer Cachexia: A Prospective, Multicenter Real World Study of a Large Cohort of Chinese Patients
Brief Title: A Multicenter Real World Study of Kanglaite for Cancer Cachexia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang Kanglaite Pharmaceutical Co.Ltd (Other)
Collaborators: NanJing PLA 81 Hospital (Other); LinkDoc Technology (Beijing) Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KLT-2018
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Cancer Cachexia
Keywords: Kanglaita Injection/Capsule; Cancer cachexia; Real-world evidences; Overall survival
MeSH Terms: interventions — kang-lai-te; Capsules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kanglaite Injection/Capsules: Kanglaite injection 200ml, iv. gtt qd×7d or more, followed by Kanglaite capsule 0.45g×6 tablets qid po×14d as one cycle for at least 4 cycles
  Interventions: Drug: Kanglaite Injection/Capsules

INTERVENTIONS:
Drug: Kanglaite Injection/Capsules — Kanglaite injection 200 mL, iv. gtt qd×7d or more, followed by Kanglaite capsule 0.45g×6 tablets qid po×14d as one cycle for at least 4 cycles
  Other Names: Coicis oil injection, Z10970091; Coix seed oil triglyceride, 03004812Z

SUMMARY:
A prospective, multi-center real-world study of the effectiveness and safety of Kanglaita Injection/Capsule in Chinese patients with cancer cachexia

DETAILED DESCRIPTION:
This is a large national-based prospective, multi-center real-world observational study. Cancer cachexia patients scheduled for sequential treatment with Kanglaite injection and capsule between August 2018 and March 2020 at 640 participating hospitals will be recruited to evaluate the effectiveness and safety of Kanglaite.

ELIGIBILITY:
Inclusion Criteria:

Patients with pathological or cytological diagnosis of lung, liver, pancreatic or stomach cancer; Patients scheduled to receive Kanglaite injection for 7 or more days, followed by Kanglaite capsule for 14 or more days; Patients willing to participate in this study and provide written informed consent.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients meeting international diagnostic criteria for cachexia:
  1. Weight loss > 5% over past 6 months or
  2. BMI<20 kg/m2 and weight loss > 2% or
  3. Sarcopenia and weight loss >2%;
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2018-08-20 (Estimated); Primary Completion 2020-03-20 (Estimated); Study Completion 2020-07-20 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2018 - 2020
  Overall survival

SECONDARY OUTCOMES:
Lean body mass | 2018 - 2020
  Lean body mass
Body weight | 2018 - 2020
  Body weight
Grade of cachexia | 2018 - 2020
  Grade of cachexia
European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire QLQ-C30 | 2018 - 2020
  European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire QLQ-C30: 30 items, including functioning, symptoms, and overall health. min: 0, max: 100. The higher values indicate higher level of functioning and quality of life
Karnofsky performance status | 2018 - 2020
  Karnofsky performance status
Patient-generated subjective global assessment (PG-SGA) | 2018 - 2020
  Patient-generated subjective global assessment (PG-SGA)
Numeric rating scale for pain | 2018 - 2020
  Numeric rating scale for pain min: 0; max: 10. The higher values indicate worse pain.
Numeric rating scale for appetite | 2018 - 2020
  Numeric rating scale for appetite min: 0; max: 10. The higher values indicate worse appetite
Synergistic antitumor effect: Overall response rate | 2018 - 2020
  Synergistic antitumor effect: Overall response rate
Synergistic antitumor effect: Disease control rate | 2018 - 2020
  Synergistic antitumor effect: Disease control rate

OTHER OUTCOMES:
Adverse events | 2018 - 2020
  Adverse events
Serious adverse event | 2018 - 2020
  Serious adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Shukui Qin, MD, Principal Investigator — NanJing PLA 81 Hospital
Locations (2):
- China (2):
  - Peking University International Hospital, Beijing, Beijing Municipality
  - NanJing PLA 81 Hospital, Nanjing, Jiangsu